CLINICAL TRIAL: NCT00855738
Title: Liceo Study: A Prospective, Observational Study On The Effectiveness Of New Antiepileptic Drugs As First Bitherapy In The Daily Clinical Practice
Brief Title: A Prospective, Observational Study On The Effectiveness Of New Antiepileptic Drugs As First Bitherapy In The Daily Clinical Practice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081144; LICEO STUDY
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2010-11

CONDITIONS: Focal Epilepsy
Keywords: epilepsy antiepileptic biotherapy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Gabapentin; Lamotrigine; Levetiracetam; Pregabalin; Tiagabine; Topiramate; Zonisamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1.0 (Other)
  Interventions: Drug: Gabapentin, Lamotrigine, Levetiracetam, Pregabalin, Oxcarbacepine, Tiagabine, Topiramate, Zonisamide

INTERVENTIONS:
Drug: Gabapentin, Lamotrigine, Levetiracetam, Pregabalin, Oxcarbacepine, Tiagabine, Topiramate, Zonisamide — * Gabapentin: up to 3.600 mg/d
  * Lamotrigine: up to 400 mg/d
  * Levetiracetam: up to 3.000 mg/d
  * Pregabalin: up to 600 mg/d
  * Oxcarbazepine: up to 2.400 mg/d
  * Tiagabine: up to 30 mg/d
  * Topiramate: up to 400 mg/d
  * Zonisamide: up to 500 mg/d
  Other Names: Neurontin, Lamictal, Lyrica, Keppra, Topamax, Gabatril, Episen, Zonegran

SUMMARY:
Assessment of the efficacy under daily clinical conditions of the new antiepileptic drugs (AEDs) gabapentin, lamotrigine, levetiracetam, oxcarbazepine, pregabalin, tiagabine and topiramate, used as first-choice combination therapy (bitherapy) in patients with focal epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Diagnosis of focal epilepsy.
* Previous failure of one or more AEDs used in monotherapy.
* Background treatment with an antiepileptic drug.
* The investigator has considered that the patient must start treatment with some of the seven new AEDs in combination therapy: lamotrigine, levetiracetam, gabapentin, oxcarbazepine, pregabalin, tiagabine and/or topiramate.
* History of seizures in the patient in the past 3 months.
* The patient or legal guardian must be able to understand the characteristics of the study and fill in the seizure diaries.
* Written informed consent.

Exclusion Criteria:

* Inability to comply with the study requirements.
* Diagnosis of generalized epilepsy or inability to establish if focal or generalized.
* Presence of serious or uncontrolled systemic disease, serious psychiatric disease or progressive neurological disease.
* History of alcoholism, drug addiction, or abuse of medicines in the past two years.
* Psychogenic seizures in the two years prior to inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081144&StudyName=A%20Prospective%2C%20Observational%20Study%20On%20The%20Effectiveness%20Of%20New%20Antiepileptic%20Drugs%20As%20First%20Bitherapy%20In%20The%20Daily%20Clinical%20Practice

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Given the observational nature of the study, the selection of treatment and dose of study medication was independent from participation in the study and was determined by daily clinical practice.
Groups:
- All Antiepileptic Drugs: Pregabalin, Levetiracetam, Topiramate, Lamotrigine, Oxcarbazepine, Zonisamide, Gabapentin: treatment, dose and frequency of administration determined by daily clinical practice
Period: Overall Study
Arm/Group | All Antiepileptic Drugs
Started | 111
At Least 1 Dose and 1 Endpoint | 108 (Received at least 1 dose of study drug and had data for at least 1 efficacy endpoint.)
Completed | 106
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1
Not completed — Subject Defaulted | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Classified as Responders
Description: Responder = decrease in number of seizures by >=50 percent (%) during the last 3 months of treatment before discontinuation (assessed at Month 3 and Month 6) versus the number of seizures that occurred during the 3 months before the baseline visit (baseline).
Time Frame: Baseline, Month 3, Month 6 (last 3 months of treatment)
Population: Full Analysis Set (FAS): intent-to-treat population = those who took at least 1 dose of study medication and had post-baseline data for at least 1 efficacy endpoint. Last Observation Carried Forward (LOCF) captures last 3 months of treatment for subjects who discontinued between Month 3 and Month 6 only. N=number of subjects with evaluable data.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 90
percent of participants
  Month 3 | 76.7 [66.6 to 84.9]
  Month 6 | 80.0 [70.2 to 87.7]
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Month 3: p-value versus baseline; Test type: Superiority or Other; p < 0.0001, McNemar
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Month 6: p-value versus baseline; Test type: Superiority or Other; p < 0.0001, McNemar

2. Secondary Outcome: Percent of Participants With Reduction in Number of Seizures >=25% and >=75% During the Last 3 Months of Treatment
Description: Percent of participants with reduction in number of seizures >=25% and >=75% during the last 3 months of treatment before discontinuation (assessed at Month 3 and Month 6) versus the 3 month period before the baseline visit.
Time Frame: Baseline, Month 3, Month 6 (last 3 months of treatment)
Population: FAS; LOCF. N=number of subjects with evaluable data.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 90
percent of participants
  Month 3: >=25% | 86.7 [77.9 to 92.9]
  Month 3: >=75% | 27.8 [18.8 to 38.2]
  Month 6: >= 25% | 86.7 [77.9 to 92.9]
  Month 6: >=75% | 54.4 [43.6 to 65.0]
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Month 3 >=25% reduction: p-value versus baseline; Test type: Superiority or Other; p < 0.0001, McNemar
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Month 3 >=75% reduction: p-value versus baseline; Test type: Superiority or Other; p < 0.0001, McNemar
Statistical Analysis 3: Comparison: All Antiepileptic Drugs; Month 6: >=25% reduction: p-value versus baseline; Test type: Superiority or Other; p < 0.0001, McNemar
Statistical Analysis 4: Comparison: All Antiepileptic Drugs; Month 6: >=75% reduction: p-value versus baseline; Test type: Superiority or Other; p < 0.0001, McNemar

3. Secondary Outcome: Percent of Seizure-free Participants During the Last 3 Months Before Discontinuation
Time Frame: Baseline, Month 3, Month 6 (last 3 months of treatment)
Population: FAS; LOCF. N=number of subjects with evaluable data.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 90
percent of participants
  Month 3 | 10.0 [4.7 to 18.1]
  Month 6 | 20.0 [12.3 to 29.8]
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Month 3: p-value versus baseline; Test type: Superiority or Other; p = 0.0039, McNemar
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Month 6: p-value versus baseline; Test type: Superiority or Other; p < 0.0001, McNemar

4. Secondary Outcome: Percent Change From Baseline in the Median Number of Seizures During the Last 3 Months of Treatment
Time Frame: Baseline, Month 3, Month 6 (last 3 months of treatment)
Population: FAS LOCF. N=number of subjects with evaluable data.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 90
percent change | -75.0 [-88.9 to -50.0]
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed Rank Test

5. Secondary Outcome: Percent of Days Without Crisis During the Study
Description: Crisis was defined as the total number of seizures during the study, the seizures at month 3 plus the seizures at month 6. The percent of days without crisis is number of days of study (date of last visit minus date of baseline visit) without crisis divided by number of days of study, multiplied by 100.
Time Frame: Baseline through Month 6 (or end of treatment)
Population: The percentage of days without crisis during the study was not evaluable because a diary with the daily number of crises was not collected.
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to First Seizure
Description: Number of days to first seizure after baseline.
Time Frame: Baseline to Month 6 (or end of treatment)
Population: FAS LOCF. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 79
days | 35.9 (40.2)

7. Secondary Outcome: Percent of Participants Who Continued on Study Medication to Month 6
Description: Retention rate: percent of participants who continued on study medication throughout the 6 Month period after inclusion in the study.
Time Frame: Baseline to Month 6
Population: FAS; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 108
percent of participants | 97.1

8. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Time Frame: Baseline, Month 3, Month 6
Population: FAS; LOCF. As no participants discontinued due to lack of efficacy, the time to exit analysis was not performed.
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 0

9. Secondary Outcome: Time to Discontinuation Due to Safety, Tolerability, or Treatment Compliance
Time Frame: Baseline, Month 3, Month 6
Population: FAS; LOCF. Due to the low number of participants who discontinued due to safety, tolerability or compliance with treatment, the time to exit analysis was not performed.
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 0

10. Secondary Outcome: Time to Discontinuation Due to Other Reasons
Time Frame: Baseline, Month 3, Month 6
Population: FAS; LOCF. Due to the low number of participants who discontinued due to other reasons, the time to exit analyses was not performed.
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 0

11. Secondary Outcome: Treatment Satisfaction Evaluated by Patient Global Impression of Change Visual Analog Scale (VAS)
Description: Patient Global Impression of Change VAS: subject rated instrument to measure subject's change in overall status; range from 0 (much better) to 10 (much worse).
Time Frame: Baseline, Month 3, Month 6
Population: FAS; LOCF. The scale for this endpoint was not collected and results were not analyzed as planned.
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 0

12. Secondary Outcome: Percent of Participants Reaching Monotherapy
Description: Percent of participants who started on more than one treatment (bitherapy) and reached monotherapy by end of study.
Time Frame: Baseline through Month 6 (or end of study)
Population: FAS; LOCF. N=number of participants who started on bitherapy.
Measure: Number (95% Confidence Interval); unit: percent of partipants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 105
percent of partipants | 2.9 [0.6 to 8.1]

13. Secondary Outcome: Percent of Participants That Reduced, Maintained and Increased Their Doses of New Antiepileptic Drugs (AED)
Time Frame: Baseline to Month 6 (or end of treatment)
Population: FAS; LOCF.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 108
percent of participants
  Reduced | 0.9 [0.0 to 5.1]
  Maintained | 68.5 [58.9 to 77.1]
  Increased | 30.6 [22.1 to 40.2]

14. Secondary Outcome: Percent of Participants That Reduced, Maintained and Increased the Doses of the Initial Treatment Administered in Monotherapy
Time Frame: Baseline through Month 6 (or end of treatment)
Population: FAS; LOCF. N= number of subjects with initial treatment administered as monotherapy.
Measure: Number; unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 3
percent of participants
  Reduced | 0.0
  Maintained | 100.0
  Increased | 0.0

15. Secondary Outcome: Change From Baseline to Month 6 in the Hospital Anxiety and Depression Scale (HADS)
Description: HADS: subject rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline to Month 6
Population: FAS; LOCF. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 92
scores on scale
  Depression | -0.5 (3.5)
  Anxiety | -0.6 (3.0)
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Depression domain: P-value vs baseline; Test type: Superiority or Other; p = 0.1797, t-test, 2 sided
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Anxiety domain: P-value vs baseline; Test type: Superiority or Other; p = 0.0433, t-test, 2 sided

16. Secondary Outcome: Change From Baseline to Month 6 in Quality of Life 10 Domains (QOLIE-10)
Description: QOLIE-10: 10-item questionnaire evaluates health-related quality of life in individuals with epliepsy. Comprised of 7 components: seizure worry, overall quality of life, emotional well-being, energy, cognitive functioning, medication effects (physical and mental effects), and social function (work, driving, social function). Total score rated 0 to 100; higher score = higher quality of life.
Time Frame: Baseline to Month 6
Population: FAS; LOCF. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 107
scores on scale
  Energy | 0.4 (17.8)
  Emotions (mood) | 0.7 (16.0)
  Daily activities | 0.6 (12.9)
  Mental function | 1.2 (20.8)
  Medication effects (physical/ mental) | -1.1 (14.9)
  Worry about seizures (impact of seizures) | 9.0 (21.1)
  Overall quality of life | 3.8 (17.2)
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Energy: p-value versus baseline; Test type: Superiority or Other; p = 0.8284, t-test, 2 sided
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Emotions (mood): p-value versus baseline; Test type: Superiority or Other; p = 0.6299, t-test, 2 sided
Statistical Analysis 3: Comparison: All Antiepileptic Drugs; Daily activities: p-value versus baseline; Test type: Superiority or Other; p = 0.6162, t-test, 2 sided
Statistical Analysis 4: Comparison: All Antiepileptic Drugs; Mental function: p-value versus baseline; Test type: Superiority or Other; p = 0.5609, t-test, 2 sided
Statistical Analysis 5: Comparison: All Antiepileptic Drugs; Medication effects (physical/ mental): p-value versus baseline; Test type: Superiority or Other; p = 0.4635, t-test, 2 sided
Statistical Analysis 6: Comparison: All Antiepileptic Drugs; Worry about seizures (impact of seizures): p-value versus baseline; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 7: Comparison: All Antiepileptic Drugs; Overall quality of life: p-value versus baseline; Test type: Superiority or Other; p = 0.0258, t-test, 2 sided

17. Secondary Outcome: Change From Baseline to Months 3 and 6 in Health Condition: Euro Quality of Life Scale (EQ-5D) Visual Analog Scale (VAS)
Description: Assessment of the health condition of the subjects using the EQ-5D VAS: subject rated questionnaire to assess health-related quality of life in terms of a single index value. Using the VAS subjects rated current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Month 3, Month 6
Population: FAS LOCF. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 105
scores on scale
  Month 3 | -0.4 (16.2)
  Month 6 | 1.2 (15.6)
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Month 3: p-value versus baseline; Test type: Superiority or Other; p = 0.7822, t-test, 2 sided
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Month 6: p-value versus baseline; Test type: Superiority or Other; p = 0.4471, t-test, 2 sided

18. Secondary Outcome: Change in Sleep Disturbances From Baseline to Month 6: Medical Outcomes Study Sleep Scale (MOS-SS)
Description: Subject rated instrument to assess key constructs of sleep; assesses sleep quality and quantity. Consists of a 6-item and 9-item overall sleep problems index measuring time to fall asleep and sleep duration in past 4 weeks; 5 subscales rated 1 (all the time) to 6 (none of the time): sleep disturbance, snoring, awaken short of breath, somnolence, and adequacy. Transformed scores range = 0 to 100; higher score indicates greater intensity of attribute. Two additional subscales = sleep quantity (range 0-24 hours) and optimal sleep (number of participants with optimal sleep 7-8 hours per night).
Time Frame: Baseline to Month 6
Population: FAS LOCF. Change from baseline in Optimal sleep is not shown as changes from baseline were only evaluated for continuous parameters. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 107
scores on scale
  Sleep disturbance | -1.7 (15.1)
  Snoring | 0.0 (15.6)
  Awake short of breath | 1.1 (14.6)
  Quantity | 0.2 (0.8)
  Adequacy | 2.8 (15.0)
  Somnolence | 0.6 (11.0)
  Sleep problems (summary 6) | -0.9 (11.7)
  Sleep problems (summary 9) | -0.9 (13.2)
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Sleep disturbance: p-value versus baseline; Test type: Superiority or Other; p = 0.2452, t-test, 2 sided
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Snoring: p-value verus baseline; Test type: Superiority or Other; p = 1.0000, t-test, 2 sided
Statistical Analysis 3: Comparison: All Antiepileptic Drugs; Awake short of breath: p-value versus baseline; Test type: Superiority or Other; p = 0.4253, t-test, 2 sided
Statistical Analysis 4: Comparison: All Antiepileptic Drugs; Quantity: p-value versus baseline; Test type: Superiority or Other; p = 0.0572, t-test, 2 sided
Statistical Analysis 5: Comparison: All Antiepileptic Drugs; Adequacy: p-value versus baseline; Test type: Superiority or Other; p = 0.0625, t-test, 2 sided
Statistical Analysis 6: Comparison: All Antiepileptic Drugs; Somnolence: p-value versus baseline; Test type: Superiority or Other; p = 0.5540, t-test, 2 sided
Statistical Analysis 7: Comparison: All Antiepileptic Drugs; Sleep problems (summary 6): p-value versus baseline; Test type: Superiority or Other; p = 0.4204, t-test, 2 sided
Statistical Analysis 8: Comparison: All Antiepileptic Drugs; Sleep problems (summary 9): p-value versus baseline; Test type: Superiority or Other; p = 0.4869, t-test, 2 sided

19. Secondary Outcome: Percent of Participants Indicating Optimal Sleep on the Optimal Sleep Subscale: Medical Outcomes Study Sleep Scale (MOS-SS)
Description: MOS-SS: subject rated instrument used to assess the key constructs of sleep; assesses sleep quantity and quality and is comprised of 12 items yielding 7 subscale scores and 2 composite index scores. Optimal sleep subscale is derived from sleep quantity average hours of sleep over the past 4 weeks; percent of participants with response YES (optimal) if sleep quantilty was 7-8 hours of sleep per night.
Time Frame: Baseline, Month 6
Population: FAS; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 108
percent of participants
  Baseline | 56.5
  Month 6 | 65.7
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Month 6: p-value versus baseline; Test type: Superiority or Other; p = 0.0863, McNemar

20. Secondary Outcome: Change From Baseline to Month 6 in Visits to a Specialist or the Emergency Room Because of Epilepsy
Description: Numerical assessment of change in the number of visits to a specialist or the emergency room because of epilepsy needed during the study.
Time Frame: Baseline to Month 6
Population: FAS; LOCF. Costs involved in health and non-health resources needed during the study were not analyzed as planned with this endpoint. N=number of subjects with visits to a specialist because of epilepsy.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 108
visits
  Number of visits to a specialist (n=94) | -0.6 (2.3)
  Number of visits to the emergency room (n=79) | -0.3 (0.9)
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Number of visits to a specialist because of epilepsy: p-value versus baseline; Test type: Superiority or Other; p = 0.0226, t-test, 2 sided
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Number of visits to the emergency room because of epilepsy: p-value versus baseline; Test type: Superiority or Other; p = 0.0017, t-test, 2 sided

21. Secondary Outcome: Change From Baseline to Month 6 in Total Number of Days Hospitalized Because of Epilepsy
Description: Numerical assessment of change in total number of days hospitalized because of epilepsy during the study.
Time Frame: Baseline to Month 6
Population: FAS; LOCF. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 76
Days | -8.0 (68.6)
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; P-value versus baseline; Test type: Superiority or Other; p = 0.3141, t-test, 2 sided

22. Secondary Outcome: Percent of Participants With Cessation of Occupation, Requirement of Caregiver, or Admission to Intensive Care Unit
Description: Percent of participants with cessation of usual occupation, requirement of an informal caregiver, and who required admission to the intensive care unit (ICU).
Time Frame: Month 6
Population: FAS; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | All Antiepileptic Drugs
Number analyzed (Participants) | 108
percent of participants
  Stopped Usual Occupation | 16.2
  Required Informal Caregiver | 6.6
  Required Admission to ICU | 0.0
Statistical Analysis 1: Comparison: All Antiepileptic Drugs; Cessation of usual occupation: p-value versus baseline; Test type: Superiority or Other; p = 0.0708, t-test, 2 sided
Statistical Analysis 2: Comparison: All Antiepileptic Drugs; Requirement of informal caregiver: p-value versus baseline; Test type: Superiority or Other; p = 1.0000, t-test, 2 sided
Statistical Analysis 3: Comparison: All Antiepileptic Drugs; Required admission to ICU: p-value versus baseline; Test type: Superiority or Other; p = 1.0000, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Includes data from baseline to 7 days after last dose of study drug.
Description: Safety Population: subjects known to have taken at least one dose of study medication.
Groups:
- All Antiepileptic Drugs (Including Pregabalin): Pregabalin, Levetiracetam, Topiramate, Lamotrigine, Oxcarbazepine, Zonisamide, Gabapentin
Arm/Group | All Antiepileptic Drugs (Including Pregabalin) | Pregabalin (Pregabalin Only)
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/40
Other Adverse Events (participants affected / at risk) | 7/111 | 5/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Antiepileptic Drugs (Including Pregabalin) (N=111) | Pregabalin (Pregabalin Only) (N=40)
Asthenia (General disorders) | 1 | 0
Weight increased (Investigations) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 4 | 3

LIMITATIONS AND CAVEATS:
This study was cancelled with 111 patients enrolled due to lack of recruitment, and inability to analyze the study by treatment groups. Seizures were analyzed by 3 month data instead of 2 month data as originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.